CLINICAL TRIAL: NCT03698474
Title: Comparison of Efficiency and Tolerance of Sodium Picosulphate/ Magnesium Citrate, Polyethylene Glycol/Ascorbate and Oral Sulfate Solution Before Colonoscopy
Brief Title: Comparison of Different Low Volume Solutions Prior to Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN102018
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-10

CONDITIONS: Colonoscopy
MeSH Terms: interventions — magnesium citrate; Polyethylene Glycols; Ascorbic Acid; Potassium, Dietary; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SPMC-S (Active Comparator): Natrium picosulfate /Magnesium citrate ( Picoprep™, oral solution) 2L in the evening before colonoscopy
  Interventions: Drug: Natrium picosulfate / Magnesium citrate
- SPMC-D (Active Comparator): Natrium picosulfate/ Magnesium citrate ( Picoprep™, oral solution) 1L in the evening and 1L in the morning before colonoscopy
  Interventions: Drug: Natrium picosulfate / Magnesium citrate
- PEGA-S (Active Comparator): Polyethylene glycol / Ascorbic acid ( Moviprep™, oral solution) 2L in the evening before colonoscopy
  Interventions: Drug: Polyethylene glycol / Ascorbic acid
- PEGA-D (Active Comparator): Polyethylene glycol / Ascorbic acid (Moviprep™, oral solution) 1L in the evening and 1L in the morning before colonoscopy
  Interventions: Drug: Polyethylene glycol / Ascorbic acid
- SULF-S (Active Comparator): Natrium/ Kalium/ Magnesium sulfate ( Eziclen™, oral solution) 1 L in the evening before colonoscopy
  Interventions: Drug: Natrium/ Kalium/ Magnesium sulfate
- SULF-D (Active Comparator): Natrium/ Kalium/ Magnesium sulfate ( Eziclen™, oral solution) 0,5 L in the evening and 0,5L in the morning before colonoscopy
  Interventions: Drug: Natrium/ Kalium/ Magnesium sulfate

INTERVENTIONS:
Drug: Natrium picosulfate / Magnesium citrate — bowel preparation formula
  Arms: SPMC-D; SPMC-S
Drug: Polyethylene glycol / Ascorbic acid — bowel preparation formula
  Arms: PEGA-D; PEGA-S
Drug: Natrium/ Kalium/ Magnesium sulfate — bowel preparation formula
  Arms: SULF-D; SULF-S

SUMMARY:
Study evaluates the head -to-head efficacy and tolerability of low volume preparations prior to colonoscopy

DETAILED DESCRIPTION:
Aim of the study: To compare the efficacy and tolerance of sodium picosulphate/magnesium citrate, polyethylene glycol/ascorbic acid and oral sulfate formula in a single or split dose regimen prior to colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* subjects referred to diagnostic or therapeutic colonoscopy

Exclusion Criteria:

* known or suspected bowel obstruction
* active bowel inflammation
* pregnancy
* prior bowel resection
* any presence of serious medical conditions ( cardiac, renal, liver disease)
* inability to obtain valid data from subject
* active bowel bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Satisfactory bowel preparation quality (Aronchick score 1-2) | one day
  Aronchick scale (1 -5)

SECONDARY OUTCOMES:
Bowel preparation tolerance assessed by Visual Analogue Scale (VAS) | one day
  VAS scale 0-10 ( 0- the best, 10 - the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kojecky, Principal Investigator — KNTB Zlin
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No